CLINICAL TRIAL: NCT01515787
Title: A Phase II/III Trial of Neoadjuvant FOLFOX With Selective Use of Combined Modality Chemoradiation Versus Preoperative Combined Modality Chemoradiation for Locally Advanced Rectal Cancer Patients Undergoing Low Anterior Resection With Total Mesorectal Excision (PROSPECT)
Brief Title: PROSPECT: Chemotherapy Alone or Chemotherapy Plus Radiation Therapy in Treating Patients With Locally Advanced Rectal Cancer Undergoing Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N1048; CDR0000715321 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-00234 (Registry Identifier: CTRP (Clinical Trials Reporting System)); U10CA031946 (NIH)
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer
Keywords: stage IIA rectal cancer; stage IIIA rectal cancer; stage IIIB rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Drug Therapy; Chemoradiotherapy; Surgical Procedures, Operative; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Patients will receive FOLFOX chemotherapy once every two weeks for 6 cycles total over a period of 12 weeks. After completing FOLFOX chemotherapy, the patient will have an MRI scan or endorectal ultrasound (ERUS) to examine the tumor. If the tumor has not decreased in size by at least 20%, the patient will receive 5FUCMT (radiation with chemotherapy). If the tumor has decreased in size by 20%, then the patient will proceed directly to surgery.
  If all borders of the tumor are normal post surgery, then the patient receives six additional cycles of FOLFOX chemotherapy. If all borders of the tumor are not normal then the patient receives chemoradiation therapy for 5.5 weeks after surgery. After chemoradiation, additional cycles of FOLFOX or similar chemotherapy will be recommended for 4 cycles or 8 weeks. Patient observation with follow up evaluations and event monitoring will occur up to 8 years post randomization.
  Interventions: Drug: FOLFOX (chemotherapy); Other: 5 FUCMT (chemoradiation); Procedure: surgery; Procedure: magnetic resonance imaging or endorectal ultrasound
- Group 2 (Active Comparator): Patients receive 5FUCMT including chemotherapy and radiation therapy for 5.5 weeks. Patients will be given either 5-fluorouracil or capecitabine and radiation therapy. After the chemoradiation therapy is completed, patients will proceed directly to surgery. Post-surgery, patients will receive FOLFOX chemotherapy once every two weeks for 8 cycles total over a period of 16 weeks. Patient observation with follow up evaluations and event monitoring will occur up to 8 years post randomization.
  Interventions: Drug: FOLFOX (chemotherapy); Other: 5 FUCMT (chemoradiation); Procedure: surgery

INTERVENTIONS:
Drug: FOLFOX (chemotherapy) — Oxaliplatin 85 mg/m^2 IV over 2 hours on day 1, leucovorin 400 mg/m^2 bolus IV over 2 hours on day 1 and 5-fluorouracil 400 mg/m^2 bolus over 5-15 minutes then 2400 mg/m^2 continual over 46-48 hours total dose IV on days 1-2. The treatment schedule repeats based on the group. Dose modifications are allowed based on adverse events.
Other: 5 FUCMT (chemoradiation) — 5-fluorouracil 225 mg/m^2 per day continuous IV infusion administered concurrently with radiation therapy for 5 or 7 days per week OR capecitabine 825 mg/m^2 twice daily administered orally and concurrently with radiation therapy for 5 days per week. Dose modifications are allowed based on adverse events.
Procedure: surgery — low anterior resection with total mesorectal excision
Procedure: magnetic resonance imaging or endorectal ultrasound
  Arms: Group 1

SUMMARY:
The standard treatment for locally advanced rectal cancer involves chemotherapy and radiation, known as 5FUCMT, (the chemotherapy drugs 5-fluorouracil/capecitabine and radiation therapy) prior to surgery. Although radiation therapy to the pelvis has been a standard and important part of treatment for rectal cancer and has been shown to decrease the risk of the cancer coming back in the same area in the pelvis, some patients experience undesirable side effects from the radiation and there have been important advances in chemotherapy, surgery, and radiation which may be of benefit. The purpose of this study is to compare the effects, both good and bad, of the standard treatment of chemotherapy and radiation to chemotherapy using a combination regimen known as FOLFOX, (the drugs 5-fluorouracil (5-FU), oxaliplatin and leucovorin) and selective use of the standard treatment, depending on response to the FOLFOX. The drugs in the FOLFOX regimen are all FDA (Food and Drug Administration) approved and have been used routinely to treat patients with advanced colorectal cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a multicenter, phase II/III study. Patients are stratified according to ECOG performance status (0 or 1 vs 2) and randomized to 1 of 2 treatment regimens. Patients will receive full supportive care while on this study.

OBJECTIVES:

Primary

1. Phase II component: To assure that neoadjuvant FOLFOX followed by selective use of 5FUCMT group (Group 1) maintains the current high rate of pelvic R0 resection and is consistent with non-inferiority for time to local recurrence (TLR).
2. Phase III component: To compare neoadjuvant FOLFOX followed by selective use of 5FUCMT (Group 1) to standard 5FUCMT (Group 2) with respect to the primary endpoint of the Disease-Free Survival (DFS).

Secondary

1. To determine if the neoadjuvant FOLFOX followed by selective use of 5FUCMT (Group 1) is non-inferior to the standard group 5FUCMT (Group 2) with respect to the proportion of patients who achieve a pathologic complete response (pCR) at the time of surgical resection.
2. To determine if the neoadjuvant FOLFOX followed by selective use of 5FUCMT (Group 1) is non-inferior to the standard 5FUCMT (Group 2) with respect to overall survival.
3. To evaluate and compare the adverse event profile and surgery complications between two groups.
4. To estimate the proportion of patients in the selective group (Group 1) who receive: 1) pre-operative 5FUCMT; 2) post-operative 5FUCMT; 3) either pre- or post-operative 5FUCMT.
5. To determine if the neoadjuvant FOLFOX followed by selective use of 5FUCMT (Group 1) is non-inferior to the standard 5FUCMT (Group 2) with respect to Local Recurrence (TLR)
6. To determine if the neoadjuvant FOLFOX followed by selective use of 5FUCMT (Group 1) is non-inferior to the standard 5FUCMT (Group 2) with respect to Neoadjuvant Response Score (NAR)

Event monitoring of patients will continue up to 8 years post randomization.

ELIGIBILITY:
Registration Inclusion Criteria:

1. Age ≥ 18 years at diagnosis
2. Diagnosis of rectal adenocarcinoma
3. Radiologically measurable or clinically evaluable disease as defined in the protocol
4. ECOG Performance Status (PS): 0, 1 or 2
5. For this patient, the standard treatment recommendation in the absence of a clinical trial would be combined modality neoadjuvant chemoradiation followed by curative intent surgical resection
6. Candidate for sphincter-sparing surgical resection prior to neoadjuvant therapy according to the primary surgeon
7. Primary surgeon is credentialed or is willing to be credentialed in Total Mesorectal Excision (TME), which entails submission of photos of a single TME specimen either before enrolling the first patient or by using the surgeon's 1st accrued case.
8. Clinical Stage: T2N1, T3N0, T3N1.

   * N2 disease is to be estimated as four or more lymph nodes that are ≥ 10 mm.
   * Clinical staging should be estimated based on the combination of the following assessments: physical exam by the primary surgeon, CT or PET/CT scan of the chest/abdomen/pelvis and either a pelvic MRI or an ultrasound (ERUS). If a pelvic MRI is peformed, it is acceptable to perform CT of the chest/abdomen, ommitting CT imaging of the pelvis.
9. The following laboratory values obtained ≤ 28 days prior to registration:

   * Absolute neutrophil count (ANC) ≥ 1500/mm^3
   * Platelet count ≥ 100,000/mm^3
   * Hemoglobin > 8.0 g/dL
   * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * SGOT (AST) ≤ 3 x ULN
   * SGPT (ALT) ≤ 3 x ULN
   * Creatinine ≤1.5 x ULN
10. Negative pregnancy test done ≤ 7 days prior to registration, for women of childbearing potential only
11. Patient of child-bearing potential is willing to employ adequate contraception
12. Provide informed written consent
13. Willing to return to enrolling medical site for all study assessments

Registration Exclusion Criteria:

1. Clinical T4 tumors
2. Primary surgeon indicates need for abdominoperineal (APR) at baseline
3. Evidence that the tumor is adherent to or invading the mesorectal fascia on imaging studies such that the surgeon would not be able to perform an R0 resection (one with negative margins)
4. Tumor is causing symptomatic bowel obstruction (patients who have had a temporary diverting ostomy are eligible).
5. Chemotherapy within 5 years prior to registration. Hormonal therapy is allowable if the disease free interval is ≥ 5 years.
6. Any prior pelvic radiation
7. Other invasive malignancy ≤ 5 years prior to registration. Exceptions are colonic polyps, non-melanoma skin cancer, ductal carcinoma in situ, bladder carcinoma in situ, or carcinoma-in-situ of the cervix.
8. Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects.

   * Pregnant women
   * Nursing women
   * Men or women of childbearing potential who are unwilling to employ adequate contraception
9. Co-morbid illnesses or other concurrent disease which, in the judgment of the clinician obtaining informed consent, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1194 (Actual)
Dates: Start 2012-06-12 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Schrag, MD, Study Chair — Dana-Farber Cancer Institute
Locations (1073):
- United States (1048):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Southern Cancer Center PC-Daphne, Daphne, Alabama
  - Southern Cancer Center PC-Mobile, Mobile, Alabama
  - Southern Cancer Center PC-Providence, Mobile, Alabama
  - Southern Cancer Center PC-Springhill, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Yuma Cancer Center, Yuma, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Highlands Oncology Group-Rogers, Rogers, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Feather River Cancer Center, Chico, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - Sutter Davis Hospital, Davis, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Sutter Cancer Research Consortium, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Northbay Cancer Center, Vacaville, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Yale-New Haven Shoreline Medical Center, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Lawrence and Memorial Cancer Center, Waterford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Hospital Cancer Institute Altamonte, Altamonte Springs, Florida
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Integrated Community Oncology Network-Southside Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network-Florida Cancer Center Beaches, Jacksonville Beach, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Florida Hospital Kissimmee, Kissimmee, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - The Watson Clinic, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - 21st Century Oncology-Orange Park, Orange Park, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Florida Urology Associates-Orlando, Orlando, Florida
  - Florida Hospital East Orlando, Orlando, Florida
  - 21st Century Oncology-Palatka, Palatka, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Integrated Community Oncology Network-Flager Cancer Center, Saint Augustine, Florida
  - Tampa General Hospital, Tampa, Florida
  - Florida Hospital Cancer Institute Winter Park, Winter Park, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Low Country Cancer Care Associates PC, Savannah, Georgia
  - Lewis Hall Singletary Oncology Center, Thomasville, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Hawaii Oncology Inc-POB I, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Presence Saint Joseph Hospital-Chicago, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Kendrick Colon and Rectal Center-Indianapolis, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Medical Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Berkshire Hematology Oncology PC, Pittsfield, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Winchester Hospital, Winchester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Beaumont Hospital - Farmington Hills, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - William Beaumont Hospital-Grosse Point, Grosse Pointe, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Lymphoma Clinic of Michigan, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Mid-Michigan Medical Center - Midland, Midland, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon and Rectal Association, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Hematology Oncology Consultants PC, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Saint Joseph Health System-Tawas City, Tawas City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Bhadresh Nayak MD PC-Warren, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Fairview Maple Grove Medical Center, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-North, Kansas City, Missouri
  - The University of Kansas Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Alpine Hematology-Oncology, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Cancer Care Specialists - Reno, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Saint Joseph Hospital, Nashua, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Southside Hospital, Bay Shore, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Huntington Hospital, Huntington, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Orange Regional Medical Center, Middletown, New York
  - NYU Winthrop Hospital, Mineola, New York
  - Mount Sinai Union Square, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Hematology Oncology Associates of Central New York-Onondaga Hill, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Carolina Surgical Clinic of Charlotte PA, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Lake Norman Hematology Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Vidant Oncology-Kenansville, Kenansville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Specialists-Matthews, Matthews, North Carolina
  - Lake Norman Hematology Oncology Specialists-Mooresville, Mooresville, North Carolina
  - Vidant Oncology-Richlands, Richlands, North Carolina
  - Carolina Oncology Associates PA, Salisbury, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Pointe, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - The Regional Cancer Center, Erie, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Armstrong Center for Medicine and Health, Kittanning, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - Drexel University School of Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Abington Memorial Hospital-Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Greenville Health System Cancer Institute-Laurens, Clinton, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - The Methodist Hospital System, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - MD Anderson Regional Care Center-Katy, Houston, Texas
  - MD Anderson Regional Care Center-Bay Area, Nassau Bay, Texas
  - MD Anderson Regional Care Center-Sugar Land, Sugar Land, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - MD Anderson Regional Care Center-The Woodlands, The Woodlands, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Sentara Martha Jefferson Hospital, Charlottesville, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Centra Lynchburg Hematology-Oncology Clinic Inc, Lynchburg, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Sentara Leigh Hospital, Norfolk, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Tri-Cities Cancer Center, Kennewick, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Seattle Cancer Care Alliance at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Spokane Valley Cancer Center-Mayfair, Spokane, Washington
  - Cancer Care Northwest-Valley, Spokane, Washington
  - Spokane Valley Cancer Center-Mission, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood North Cancer Treatment Center, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center - Eau Claire, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System Eau Claire Hospital-Luther Campus, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Saint Clare's Hospital, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (16):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - London Regional Cancer Program, London, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Niagara Health System-Saint Catharines General, Saint Catharines, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - PEI Cancer Treatment Centre-Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - McGill University Department of Oncology, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Shaare Zedek Medical Center, Jerusalem, Israel
- Switzerland (8):
  - Kantonsspital Aarau, Aarau
  - University Hospital Basel, Basel
  - Oncology Institute of Southern Switzerland, Bellinzona
  - Kantonsspital Graubunden, Chur
  - University Hospital of Lausanne, Lausanne
  - Kantonsspital Winterthur, Winterthur
  - Zurich Im Park, Zurich
  - Zurich Hirslanden Klinik, Zurich

REFERENCES:
- [Derived] Zhang T, Shi L, Jian L, Jiang J, Qiu Y, Xie F, Zhang J, Peng H, Zhong L, Chen Y, Zhong Y, Deng Y; FOWARC Group. Clinical Benefit and Cost-Effectiveness of FOLFOX Versus LCCRT in Neoadjuvant Treatment for Patients with Locally Advanced Rectal Cancer: An Economic Analysis of the FOWARC and PROSPECT Trial. Ann Surg Oncol. 2025 Dec 11. doi: 10.1245/s10434-025-18802-8. Online ahead of print. PMID 41379261
- [Derived] Felder S, Frakes J, George M, Rosen A, Sahin IH. Which Treatment for Which Patient: Rectal Cancer Management After PROSPECT Trial. Oncology (Williston Park). 2024 May 13;38(5):187-190. doi: 10.46883/2024.25921019. PMID 38776515
- [Derived] Schrag D, Shi Q, Weiser MR, Gollub MJ, Saltz LB, Musher BL, Goldberg J, Al Baghdadi T, Goodman KA, McWilliams RR, Farma JM, George TJ, Kennecke HF, Shergill A, Montemurro M, Nelson GD, Colgrove B, Gordon V, Venook AP, O'Reilly EM, Meyerhardt JA, Dueck AC, Basch E, Chang GJ, Mamon HJ. Preoperative Treatment of Locally Advanced Rectal Cancer. N Engl J Med. 2023 Jul 27;389(4):322-334. doi: 10.1056/NEJMoa2303269. Epub 2023 Jun 4. PMID 37272534
- [Derived] Basch E, Dueck AC, Mitchell SA, Mamon H, Weiser M, Saltz L, Gollub M, Rogak L, Ginos B, Mazza GL, Colgrove B, Chang G, Minasian L, Denicoff A, Thanarajasingam G, Musher B, George T, Venook A, Farma J, O'Reilly E, Meyerhardt JA, Shi Q, Schrag D. Patient-Reported Outcomes During and After Treatment for Locally Advanced Rectal Cancer in the PROSPECT Trial (Alliance N1048). J Clin Oncol. 2023 Jul 20;41(21):3724-3734. doi: 10.1200/JCO.23.00903. Epub 2023 Jun 4. PMID 37270691
- [Derived] Schrag D, Weiser M, Saltz L, Mamon H, Gollub M, Basch E, Venook A, Shi Q. Challenges and solutions in the design and execution of the PROSPECT Phase II/III neoadjuvant rectal cancer trial (NCCTG N1048/Alliance). Clin Trials. 2019 Apr;16(2):165-175. doi: 10.1177/1740774518824539. Epub 2019 Jan 28. PMID 30688523
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://www.cancer.gov/about-cancer/treatment/clinical-trials/search/v?id=NCI-2012-00234&q=N1048

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Patients will receive FOLFOX chemotherapy once every two weeks for 6 cycles total over a period of 12 weeks. After completing FOLFOX chemotherapy, the patient will have an MRI scan or endorectal ultrasound (ERUS) to examine the tumor. If the tumor has not decreased in size by at least 20%, the patient will receive 5FUCMT (radiation with chemotherapy). If the tumor has decreased in size by 20%, then the patient will proceed directly to surgery. >
  > If all borders of the tumor are normal post surgery, then the patient receives six additional cycles of FOLFOX chemotherapy. If all borders of the tumor are not normal then the patient receives chemoradiation therapy for 5.5 weeks after surgery. After chemoradiation, additional cycles of FOLFOX or similar chemotherapy will be recommended for 4 cycles or 8 weeks.>
  > FOLFOX (chemotherapy): Oxaliplatin 85 mg/m^2 IV over 2 hours on day 1, leucovorin 400 mg/m^2 bolus IV over 2 hours on day 1 and 5-fluorouracil 400 mg/m^2 bolus over 5-15 minutes then 2400 mg/m^2 continual over 46-48 hours total dose IV on days 1-2. The treatment schedule repeats based on the group.>
  > 5 FUCMT (chemoradiation): 5-fluorouracil 225 mg/m^2 per day continuous IV infusion administered concurrently with radiation therapy for 5 or 7 days per week OR capecitabine 825 mg/m^2 twice daily administered orally and concurrently with radiation therapy for 5 days per week.
- Group 2: Patients receive 5FUCMT including chemotherapy and radiation therapy for 5.5 weeks. Patients will be given either 5-fluorouracil or capecitabine and radiation therapy. After the chemoradiation therapy is completed, patients will proceed directly to surgery. Post-surgery, patients will receive FOLFOX chemotherapy once every two weeks for 8 cycles total over a period of 16 weeks. Patient observation with follow up evaluations and event monitoring will occur up to 8 years post randomization.>
  > FOLFOX (chemotherapy): Oxaliplatin 85 mg/m^2 IV over 2 hours on day 1, leucovorin 400 mg/m^2 bolus IV over 2 hours on day 1 and 5-fluorouracil 400 mg/m^2 bolus over 5-15 minutes then 2400 mg/m^2 continual over 46-48 hours total dose IV on days 1-2. The treatment schedule repeats based on the group. Dose modifications are allowed based on adverse events.>
  > 5 FUCMT (chemoradiation): 5-fluorouracil 225 mg/m^2 per day continuous IV infusion administered concurrently with radiation therapy for 5 or 7 days per week OR capecitabine 825 mg/m^2 twice daily administered orally and concurrently with radiation therapy for 5 days per week. Dose modifications are allowed based on adverse events.>
  > surgery: low anterior resection with total mesorectal excision
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 597 | 597
Completed | 585 | 543
Not Completed | 12 | 54

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Patients will receive FOLFOX chemotherapy once every two weeks for 6 cycles total over a period of 12 weeks. After completing FOLFOX chemotherapy, the patient will have an MRI scan or endorectal ultrasound (ERUS) to examine the tumor. If the tumor has not decreased in size by at least 20%, the patient will receive 5FUCMT (radiation with chemotherapy). If the tumor has decreased in size by 20%, then the patient will proceed directly to surgery. >
  > If all borders of the tumor are normal post surgery, then the patient receives six additional cycles of FOLFOX chemotherapy. If all borders of the tumor are not normal then the patient receives chemoradiation therapy for 5.5 weeks after surgery. After chemoradiation, additional cycles of FOLFOX or similar chemotherapy will be recommended for 4 cycles or 8 weeks. >
  > FOLFOX (chemotherapy): Oxaliplatin 85 mg/m^2 IV over 2 hours on day 1, leucovorin 400 mg/m^2 bolus IV over 2 hours on day 1 and 5-fluorouracil 400 mg/m^2 bolus over 5-15 minutes then 2400 mg/m^2 continual over 46-48 hours total dose IV on days 1-2. The treatment schedule repeats based on the group. >
  > 5 FUCMT (chemoradiation): 5-fluorouracil 225 mg/m^2 per day continuous IV infusion administered concurrently with radiation therapy for 5 or 7 days per week OR capecitabine 825 mg/m^2 twice daily administered orally and concurrently with radiation therapy for 5 days per week.
- Group 2: Patients receive 5FUCMT including chemotherapy and radiation therapy for 5.5 weeks. Patients will be given either 5-fluorouracil or capecitabine and radiation therapy. After the chemoradiation therapy is completed, patients will proceed directly to surgery. Post-surgery, patients will receive FOLFOX chemotherapy once every two weeks for 8 cycles total over a period of 16 weeks. >
  > FOLFOX (chemotherapy): Oxaliplatin 85 mg/m^2 IV over 2 hours on day 1, leucovorin 400 mg/m^2 bolus IV over 2 hours on day 1 and 5-fluorouracil 400 mg/m^2 bolus over 5-15 minutes then 2400 mg/m^2 continual over 46-48 hours total dose IV on days 1-2. The treatment schedule repeats based on the group. Dose modifications are allowed based on adverse events.>
  > 5 FUCMT (chemoradiation): 5-fluorouracil 225 mg/m^2 per day continuous IV infusion administered concurrently with radiation therapy for 5 or 7 days per week OR capecitabine 825 mg/m^2 twice daily administered orally and concurrently with radiation therapy for 5 days per week. Dose modifications are allowed based on adverse events.>
  > surgery: low anterior resection with total mesorectal excision
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 585 | 543 | 1128
Age, Continuous [Median (Full Range); unit: years] | 57 [19 to 91] | 57 [25 to 84] | 57 [19 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 173 | 389
  Male | 369 | 370 | 739
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 48 | 96
  Not Hispanic or Latino | 516 | 475 | 991
  Unknown or Not Reported | 21 | 20 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 31 | 19 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 17 | 49
  White | 492 | 467 | 959
  More than one race | 30 | 40 | 70
  Unknown or Not Reported | 0 | 0 | 0
Country of residence [Count of Participants; unit: Participants]
  Canada | 51 | 45 | 96
  Switzerland | 10 | 9 | 19
  United States | 524 | 489 | 1013
Body-mass index [Median (Full Range); unit: kg/m^2] | 28.4 [14.5 to 65.4] | 28.1 [15.8 to 81.4] | 28.3 [14.5 to 81.4]
History of diabetes [Count of Participants; unit: Participants]
  Yes | 81 | 83 | 164
  No | 504 | 460 | 964
History of cardiovascular disease [Count of Participants; unit: Participants]
  Yes | 106 | 98 | 204
  No | 479 | 445 | 924
Highest education level [Count of Participants; unit: Participants] — Population: Missing Patient Data
  Participants
    Less than high school: number analyzed (Participants) | 568 | 531 | 1099
    Less than high school | 29 | 29 | 58
    High school diploma or GED certificate | 214 | 201 | 415
    Some college | 119 | 102 | 221
    College degree or higher | 206 | 199 | 405
ECOG performance-status score [Count of Participants; unit: Participants] — ECOG = 0: Fully active, able to carry on all pre-disease performance without restriction. > ECOG = 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. > ECOG = 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours. > ECOG = 0 is better. ECOG = 2 is worse.
  Participants
    0 or 1 | 582 | 540 | 1122
    2 | 3 | 3 | 6
Primary rectal tumor on digital examination [Count of Participants; unit: Participants] — Population: Missing Patient Data
  Participants
    Rectal tumor not palpable: number analyzed (Participants) | 580 | 536 | 1116
    Rectal tumor not palpable | 290 | 259 | 549
    Rectal tumor palpable | 290 | 277 | 567
Rectal tumor location [Median (Full Range); unit: cm] | 8 [2 to 25] | 8 [2 to 18] | 8 [2 to 25]
Rectal tumor location [Count of Participants; unit: Participants]
  ≤5 cm from anal verge | 83 | 89 | 172
  >5 to ≤10 cm from anal verge | 375 | 344 | 719
  >10 cm from anal verge | 127 | 109 | 236
Clinical stage [Count of Participants; unit: Participants] — Population: T1 is if the maximum pre-biopsy diameter was ≤ 2 cm and had at most one of the following high-risk features: poorly differentiated histology, location on the mucosal (non-hair bearing) lip or ear, presence of perineural invasion, or depth of invasion to Clark's level ≥ IV or > 2 mm.T2 is if > 2 cm in maximum pre-biopsy diameter or had ≥ 2 of the 7th edition AJCC high-risk features. T3 is if invaded the one or more of the facial bones (including the maxilla, mandible, orbit, or temporal bones.
  Participants
    T2 node positive: number analyzed (Participants) | 584 | 543 | 1127
    T2 node positive | 63 | 38 | 101
    T3 node negative | 232 | 198 | 430
    T3 node positive | 289 | 307 | 596
Staging performed with MRI [Count of Participants; unit: Participants]
  Yes | 494 | 458 | 952
  No | 91 | 85 | 176

OUTCOME MEASURES:

1. Primary Outcome: Pelvic R0 Resection Rate
Description: Number of Participants with Pelvic R0 Resection
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Patients will receive FOLFOX chemotherapy once every two weeks for 6 cycles total over a period of 12 weeks. After completing FOLFOX chemotherapy, the patient will have an MRI scan or endorectal ultrasound (ERUS) to examine the tumor. If the tumor has not decreased in size by at least 20%, the patient will receive 5FUCMT (radiation with chemotherapy). If the tumor has decreased in size by 20%, then the patient will proceed directly to surgery.
  >
  > If all borders of the tumor are normal post surgery, then the patient receives six additional cycles of FOLFOX chemotherapy. If all borders of the tumor are not normal then the patient receives chemoradiation therapy for 5.5 weeks after surgery. After chemoradiation, additional cycles of FOLFOX or similar chemotherapy will be recommended for 4 cycles or 8 weeks.
  >
  > FOLFOX (chemotherapy): Oxaliplatin 85 mg/m^2 IV over 2 hours on day 1, leucovorin 400 mg/m^2 bolus IV over 2 hours on day 1 and 5-fluorouracil 400 mg/m^2 bolus over 5-15 minutes then 2400 mg/m^2 continual over 46-48 hours total dose IV on days 1-2. The treatment schedule repeats based on the group.
  * FUCMT (chemoradiation): 5-fluorouracil 225 mg/m^2 per day continuous IV infusion administered concurrently with radiation therapy for 5 or 7 days per week OR capecitabine 825 mg/m^2 twice daily administered orally and concurrently with radiation therapy for 5 days per week.
- Group 2: Patients receive 5FUCMT including chemotherapy and radiation therapy for 5.5 weeks. Patients will be given either 5-fluorouracil or capecitabine and radiation therapy. After the chemoradiation therapy is completed, patients will proceed directly to surgery. Post-surgery, patients will receive FOLFOX chemotherapy once every two weeks for 8 cycles total over a period of 16 weeks. Patient observation with follow up evaluations and event monitoring will occur up to 8 years post randomization.
  >
  > FOLFOX (chemotherapy): Oxaliplatin 85 mg/m^2 IV over 2 hours on day 1, leucovorin 400 mg/m^2 bolus IV over 2 hours on day 1 and 5-fluorouracil 400 mg/m^2 bolus over 5-15 minutes then 2400 mg/m^2 continual over 46-48 hours total dose IV on days 1-2. The treatment schedule repeats based on the group. Dose modifications are allowed based on adverse events.
  >
  > 5 FUCMT (chemoradiation): 5-fluorouracil 225 mg/m^2 per day continuous IV infusion administered concurrently with radiation therapy for 5 or 7 days per week OR capecitabine 825 mg/m^2 twice daily administered orally and concurrently with radiation therapy for 5 days per week. Dose modifications are allowed based on adverse events.
  >
  > surgery: low anterior resection with total mesorectal excision
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 535 | 510
Participants | 529 | 495

2. Primary Outcome: DFS
Description: Disease-free Survival (DFS): The distribution of DFS by group will be estimated using the method of Kaplan-Meier. 5 year disease free rates by treatment group with confidence intervals based on Kaplan-Meier curves will be reported. Log-rank test will be used to compare DFS between two treatment groups. Hazard ratio with confidence interval will be estimated based on Cox proportional hazard model. The Cox proportional hazard model will be used for multivariate analysis.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Group 2: Patients receive 5FUCMT including chemotherapy and radiation therapy for 5.5 weeks. Patients will be given either 5-fluorouracil or capecitabine and radiation therapy. After the chemoradiation therapy is completed, patients will proceed directly to surgery. Post-surgery, patients will receive FOLFOX chemotherapy once every two weeks for 8 cycles total over a period of 16 weeks.
  >
  > FOLFOX (chemotherapy): Oxaliplatin 85 mg/m^2 IV over 2 hours on day 1, leucovorin 400 mg/m^2 bolus IV over 2 hours on day 1 and 5-fluorouracil 400 mg/m^2 bolus over 5-15 minutes then 2400 mg/m^2 continual over 46-48 hours total dose IV on days 1-2. The treatment schedule repeats based on the group. Dose modifications are allowed based on adverse events.
  >
  > 5 FUCMT (chemoradiation): 5-fluorouracil 225 mg/m^2 per day continuous IV infusion administered concurrently with radiation therapy for 5 or 7 days per week OR capecitabine 825 mg/m^2 twice daily administered orally and concurrently with radiation therapy for 5 days per week. Dose modifications are allowed based on adverse events.
  >
  > surgery: low anterior resection with total mesorectal excision
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 585 | 543
Participants | 114 | 113
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Non-Inferiority — Disease recurrence or death in order to have 85% power to reject the null hypothesis. Noninferiority of the intervention could be claimed if the upper limit of the two-sided 90.2% confidence interval of the hazard ratio for disease recurrence or death did not exceed the 1.29 noninferiority margin; p = 0.005, kaplan meier; Hazard Ratio (HR) = 0.92, 90.2% CI 2-sided [0.74 to 1.14]

3. Secondary Outcome: Pathologic Complete Response
Description: Pathologic Complete Response (pCR): The pCR rate is defined as number of patients who achieve pCR divided by total number of patients included in the analysis population (see definition in Section 16.3.3.1) in each group. Patients who didn't undergo surgery will be classified as non-pCR. Point estimate and confidence interval (according to approach of Duffy and Santner) will be calculated by treatment groups. Chi-square test will be used to compare the pCR rates between groups.
Time Frame: Up to 8 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 535 | 510
Participants | 117 | 124

4. Secondary Outcome: Overall Survival
Description: Overall Survival (OS): OS is defined as time from randomization to the date of death due to all causes. The distribution of OS by group will be estimated using the method of Kaplan-Meier. Five year survival rates by treatment group with confidence intervals based on Kaplan-Meier curves will be reported. Logrank test will be used to compare OS between two treatment groups. Hazard ratio with confidence interval will be estimated based on Cox proportional hazard model. The Cox proportional hazard model will be used for multivariate analysis.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 585 | 543
Participants | 74 | 67
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority; Hazard Ratio (HR) = 1.04, 95.0% CI 2-sided [0.74 to 1.44]

5. Secondary Outcome: Rates of Receiving Pre- or Post-operative 5FUCMT
Description: Rates of Receiving 5FUCMT: For selective group patients, the proportion of patients who received 1) pre-operative 5FUCMT, 2) post-operative 5FUCMT, 3) either pre or post-operative 5FUCMT, and confidence intervals (according to approach of Duffy and Santner) will be reported.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 585 | 543
Participants | 61 | 543

6. Secondary Outcome: Local Recurrence (TLR):
Description: Time to Local Recurrence (TLR): The distribution of TLR by group will be estimated using the method of Kaplan-Meier. 5 year local recurrence free rates by treatment group with confidence intervals based on Kaplan-Meier curves will be reported. The comparison of the cumulative incidence of local recurrence between groups, treating distant recurrence and death as competing risks using the test of Gray (Annals of Statistics, 1988) will be conducted.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 585 | 543
Participants | 9 | 7
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority; Hazard Ratio (HR) = 1.18, 95.0% CI 2-sided [0.44 to 3.16]

7. Secondary Outcome: Neoadjuvant Rectal Score
Description: neoadjuvant rectal (NAR) score =[5 * pN - 3(cT - pT) + 12]^2/9.61. cT is an element of the set {1, 2, 3, 4}, pT is in {0, 1, 2, 3, 4}, and pN is in {0, 1, 2}. cT clinical tumor stage, pT pathologic tumor stage, pN pathologic nodal stage. Low (NAR <8), intermediate (NAR = 8-16), and high (NAR >16). Low is better and high is worse.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 535 | 510
Participants
  Low (< 8) | 157 | 161
  Intermediate (8-16) | 247 | 230
  High (> 16) | 130 | 114

ADVERSE EVENTS:
Time Frame: Up to 5 years
Groups:
- Group 1: 5 FUCMT (chemoradiation): 5-fluorouracil 225 mg/m^2 per day continuous IV infusion administered concurrently with radiation therapy for 5 or 7 days per week OR capecitabine 825 mg/m^2 twice daily administered orally and concurrently with radiation therapy for 5 days per week.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 74/585 | 67/543
Serious Adverse Events (participants affected / at risk) | 10/585 | 7/543
Other Adverse Events (participants affected / at risk) | 582/585 | 534/543
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=585) | Group 2 (N=543)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Rectal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 1 (1) | 2 (2)
Sudden death NOS (General disorders) | 2 (2) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=585) | Group 2 (N=543)
Anemia (Blood and lymphatic system disorders) | 74 (168) | 65 (106)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 5 (9) | 3 (4)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (13) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Spleen disorder (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 2 (2)
Asystole (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 4 (4) | 6 (7)
Chest pain - cardiac (Cardiac disorders) | 3 (4) | 4 (4)
Heart failure (Cardiac disorders) | 2 (2) | 3 (4)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Mobitz (type) II atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (4) | 2 (2)
Palpitations (Cardiac disorders) | 2 (3) | 3 (4)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 5 (6)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 7 (10)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 2 (13) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 4 (4) | 2 (5)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 3 (3)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (4)
Blurred vision (Eye disorders) | 3 (3) | 2 (3)
Dry eye (Eye disorders) | 3 (8) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 4 (8) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Optic nerve disorder (Eye disorders) | 1 (1) | 1 (2)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 1 (2) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 3 (5) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 15 (22) | 19 (22)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 3 (7) | 4 (4)
Anal mucositis (Gastrointestinal disorders) | 2 (4) | 5 (7)
Anal pain (Gastrointestinal disorders) | 3 (4) | 5 (6)
Anal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2) | 7 (9)
Colitis (Gastrointestinal disorders) | 4 (4) | 5 (5)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colonic hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 7 (8) | 5 (6)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 378 (1459) | 249 (567)
Dental caries (Gastrointestinal disorders) | 1 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 401 (1537) | 442 (1490)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 6 (8)
Dyspepsia (Gastrointestinal disorders) | 10 (19) | 6 (8)
Dysphagia (Gastrointestinal disorders) | 132 (318) | 35 (47)
Enterocolitis (Gastrointestinal disorders) | 1 (2) | 3 (4)
Esophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Esophagitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 7 (12) | 15 (22)
Flatulence (Gastrointestinal disorders) | 7 (27) | 11 (16)
Gastric fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (3) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 (18) | 2 (2)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 16 (17) | 24 (35)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 2 (3) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 6 (7) | 6 (11)
Ileal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 2 (2) | 3 (3)
Ileal stenosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 9 (9) | 12 (13)
Jejunal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 246 (647) | 119 (189)
Nausea (Gastrointestinal disorders) | 433 (1904) | 326 (727)
Oral dysesthesia (Gastrointestinal disorders) | 2 (4) | 1 (1)
Oral pain (Gastrointestinal disorders) | 4 (4) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (3)
Proctitis (Gastrointestinal disorders) | 1 (1) | 9 (12)
Rectal fistula (Gastrointestinal disorders) | 1 (1) | 3 (3)
Rectal hemorrhage (Gastrointestinal disorders) | 19 (31) | 13 (19)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 6 (7)
Rectal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 8 (9) | 12 (18)
Rectal perforation (Gastrointestinal disorders) | 2 (3) | 1 (1)
Rectal stenosis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 7 (7) | 22 (27)
Stomach pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 188 (383) | 125 (196)
Chills (General disorders) | 9 (12) | 1 (2)
Edema limbs (General disorders) | 12 (28) | 5 (10)
Fatigue (General disorders) | 534 (3408) | 455 (1605)
Fever (General disorders) | 11 (13) | 4 (5)
Gen disord and admin site conds-Oth spec (General disorders) | 11 (27) | 6 (9)
Localized edema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 2 (4) | 1 (1)
Non-cardiac chest pain (General disorders) | 4 (4) | 4 (4)
Pain (General disorders) | 405 (1514) | 410 (1202)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 2 (2)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 7 (9) | 0 (0)
Anaphylaxis (Immune system disorders) | 3 (4) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 2 (4) | 4 (4)
Anorectal infection (Infections and infestations) | 2 (2) | 1 (1)
Appendicitis (Infections and infestations) | 2 (3) | 2 (3)
Bladder infection (Infections and infestations) | 1 (1) | 2 (3)
Bone infection (Infections and infestations) | 0 (0) | 4 (4)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 2 (2) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (3) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (1)
Endocarditis infective (Infections and infestations) | 1 (1) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 10 (11) | 20 (21)
Kidney infection (Infections and infestations) | 2 (3) | 1 (1)
Lip infection (Infections and infestations) | 1 (2) | 0 (0)
Lung infection (Infections and infestations) | 3 (5) | 4 (5)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 2 (3) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (3) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 1 (1) | 3 (3)
Peritoneal infection (Infections and infestations) | 0 (0) | 4 (4)
Rash pustular (Infections and infestations) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 9 (9) | 9 (10)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 5 (7) | 5 (6)
Small intestine infection (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (3)
Stoma site infection (Infections and infestations) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 4 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 8 (9) | 9 (13)
Wound infection (Infections and infestations) | 4 (4) | 9 (9)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Biliary anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (2) | 12 (14)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 2 (3)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Gastric anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 3 (5) | 2 (3)
Intestinal stoma leak (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraoperative urinary injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Large intestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Prolapse of intestinal stoma (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
Rectal anastomotic leak (Injury, poisoning and procedural complications) | 2 (2) | 6 (7)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 5 (14) | 0 (0)
Venous injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Alanine aminotransferase increased (Investigations) | 42 (86) | 8 (13)
Alkaline phosphatase increased (Investigations) | 18 (45) | 14 (26)
Aspartate aminotransferase increased (Investigations) | 44 (99) | 10 (15)
Blood bilirubin increased (Investigations) | 6 (10) | 6 (7)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 2 (2)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1)
Cholesterol high (Investigations) | 2 (6) | 3 (5)
Creatinine increased (Investigations) | 18 (30) | 17 (23)
ECG QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
GGT increased (Investigations) | 1 (2) | 0 (0)
Hemoglobin increased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 2 (7) | 2 (2)
Investigations - Other, specify (Investigations) | 6 (16) | 4 (11)
Lipase increased (Investigations) | 1 (1) | 2 (2)
Lymphocyte count decreased (Investigations) | 21 (46) | 74 (145)
Lymphocyte count increased (Investigations) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 158 (277) | 24 (32)
Platelet count decreased (Investigations) | 61 (152) | 24 (34)
Weight gain (Investigations) | 3 (8) | 2 (6)
Weight loss (Investigations) | 23 (41) | 27 (37)
White blood cell decreased (Investigations) | 53 (120) | 37 (48)
Acidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 277 (904) | 216 (437)
Dehydration (Metabolism and nutrition disorders) | 20 (22) | 40 (52)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 41 (93) | 22 (40)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (5) | 8 (8)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 18 (39) | 19 (27)
Hypocalcemia (Metabolism and nutrition disorders) | 16 (24) | 15 (21)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 26 (34) | 28 (46)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (10) | 8 (10)
Hyponatremia (Metabolism and nutrition disorders) | 24 (38) | 26 (35)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 3 (4) | 5 (5)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (31) | 10 (24)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 6 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 (9) | 14 (20)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 (7) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 6 (9) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (9) | 3 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (4)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (6) | 0 (0)
Leukemia second to oncology chemo (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (4) | 1 (2)
Dizziness (Nervous system disorders) | 18 (29) | 12 (17)
Dysesthesia (Nervous system disorders) | 4 (13) | 0 (0)
Dysgeusia (Nervous system disorders) | 20 (49) | 12 (15)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 15 (29) | 11 (13)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 5 (10) | 4 (6)
Muscle weakness left-sided (Nervous system disorders) | 1 (1) | 0 (0)
Muscle weakness right-sided (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Oth spec (Nervous system disorders) | 4 (8) | 5 (6)
Paresthesia (Nervous system disorders) | 24 (70) | 8 (18)
Peripheral motor neuropathy (Nervous system disorders) | 5 (7) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 522 (3697) | 370 (1411)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 2 (5)
Spasticity (Nervous system disorders) | 1 (3) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 4 (4)
Syncope (Nervous system disorders) | 11 (11) | 10 (13)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 4 (15) | 0 (0)
Anxiety (Psychiatric disorders) | 276 (1215) | 201 (609)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 154 (547) | 131 (343)
Insomnia (Psychiatric disorders) | 17 (56) | 18 (31)
Irritability (Psychiatric disorders) | 1 (4) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 14 (18) | 17 (25)
Chronic kidney disease (Renal and urinary disorders) | 2 (9) | 3 (4)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 4 (4)
Hematuria (Renal and urinary disorders) | 2 (2) | 3 (3)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 6 (8) | 11 (15)
Renal calculi (Renal and urinary disorders) | 1 (1) | 3 (3)
Urinary fistula (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 6 (10) | 18 (26)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 3 (3)
Urinary retention (Renal and urinary disorders) | 5 (6) | 6 (14)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 4 (5)
Urinary tract pain (Renal and urinary disorders) | 3 (4) | 9 (14)
Urinary urgency (Renal and urinary disorders) | 3 (3) | 5 (6)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 5 (9) | 5 (9)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Prostatic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (24) | 7 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 187 (587) | 119 (251)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (29) | 3 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 3 (8) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (8)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 17 (49) | 7 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (6) | 14 (26)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 7 (12) | 15 (18)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (9) | 4 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 (13) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 (19) | 8 (9)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 8 (12) | 9 (11)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (13) | 7 (8)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (4) | 2 (5)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Social circumstances - Other, specify (Social circumstances) | 1 (5) | 0 (0)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 3 (3) | 4 (4)
Flushing (Vascular disorders) | 1 (1) | 1 (2)
Hematoma (Vascular disorders) | 3 (3) | 0 (0)
Hot flashes (Vascular disorders) | 6 (9) | 2 (2)
Hypertension (Vascular disorders) | 60 (154) | 48 (104)
Hypotension (Vascular disorders) | 19 (24) | 16 (20)
Thromboembolic event (Vascular disorders) | 20 (33) | 13 (14)
Vascular disorders - Other, specify (Vascular disorders) | 3 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT01515787/Prot_SAP_000.pdf